CLINICAL TRIAL: NCT07238608
Title: UPRISE Unravelling Ultrafine Particulate Matter and Micro Nano Plastic's Mechanisms of Impact on Fetal Health
Brief Title: Impact of UFPs and MNPs on Fetal Health
Acronym: UPRISE
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Hasselt University (Other); Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Alba Ruiz Gaitán, MD, PhD, Instituto de Investigacion Sanitaria La Fe
Other Study IDs: UPRISE; 1011566 (Other Grant/Funding Number: European Union)
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pregnant Women
Keywords: non-communicable diseases; Ultrafine Particulate; micro nano plastics
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — PBMNCs from cord blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case-control design: The study includes 1600 participants, providing a substantial sample for analysis. The focus is on newborns (age 0), making the study particularly relevant for understanding factors and outcomes related to this very early stage of life. The sex of the participants is expected to be randomly distributed. A control arm of full-term neonates (>37 weeks) will be recruited for a 1:2 ratio in Greece and Spain. ENVIRONAGE, Belgium, employs a nested case-control design, making use of its prospective cohort framework that is already in place.
- Personal Exposure Monitoring PEM Substudy: The study consists of 150 mothers, with 50 from each location. All participants are females aged over 18 years. The sex of the participants is expected to be randomly distributed.

SUMMARY:
This project aims at unravelling mechanisms by which exposure to air pollution (in particular Ultrafine Particulate (UFP, PM0.1), and micro nano plastic's) interferes with the normal foetus development, with a short-term causal effect in higher likeliness of preterm delivery which, in consequence, precondition a higher likeliness to suffer non-communicable diseases (NCD) later in the life.

DETAILED DESCRIPTION:
The characteristics of this study population are as follows:

1. Case-control design The study includes 1600 participants, providing a substantial sample for analysis. The focus is on newborns (age 0), making the study particularly relevant for understanding factors and outcomes related to this very early stage of life. The sex of the participants is expected to be randomly distributed. A control arm of full-term neonates (>37 weeks) will be recruited for a 1:2 ratio in Greece and Spain.
2. Personal Exposure Monitoring PEM Substudy:

The study consists of 150 mothers, with 50 from each location. All participants are females aged over 18 years. The sex of the participants is expected to be randomly distributed.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to sign the informed consent;
* Non-smoking mothers and no exposure to environmental (second-hand) smoke (smoking influences UFP measurements);
* ≥18 years old (mothers have to place sensors, mothers with childhood pregnancies may live at their parental home);
* Not expecting to terminate the pregnancy (no measurements of the child);
* Having resided in the geographical area of research for a minimum period of 1 year (to be eligible for modeling exposures).

Exclusion Criteria:

* First visit after 11 weeks of gestation (to ensure 2-week monitoring in the first trimester);
* Pregnancy complications that limit exposure measurements in urine (because it may cause polyuria, for example, gestational diabetes);
* Known kidney disease (might influence exposure measurements in urine);
* Multiple pregnancy (twin or more pregnancies may have a higher risk for complications or preterm birth, no measurements in the last trimester).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Pregnant mothers will be recruited at the first antenatal visit (around eight weeks of gestation).
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
PreTerm Birth | at the moment of birth
Small for Gestational Age | at the moment of birth
Low Birth Weigth | at the moment of birth

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Investigación Sanitaria La Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.uprise-horizon.eu/